CLINICAL TRIAL: NCT05288621
Title: Electroacupuncture at "Four Sacral Points" for Benigh Prosatic Hyperplasia/Lower Urinary Tract Symptoms: A Randomized Controlled Trial
Brief Title: Benigh Prosatic Hyperplasia/Lower Urinary Tract Symptoms
Acronym: BPH/LUTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jie Zhou, Deputy Chief Physician, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3rdZhejiangCMU
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms; electroacupuncture; four sacral points
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Electroacupuncture; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture at'four sacral points' (Experimental): The participants in the electroacupuncture at'four sacral points'group will receive treatment that consists of 8 acupuncture sessions over an 4-week period after baseline (2 sessions in each week), each for 30 minutes. Hua Tuo brand disposable acupunctureneedles (size 0.40 × 100mm) and electronic needle therapy instrument SDZ-IIB will be used.The device will be set at a frequency of 2.0 Hz, continuous wave and a moderate intensity the patient can tolerate. Electrostimulation will be performed for 30 min during each treatment. BL30 (Baihuanshu )(both sides and BL35 (Huiyang )(both sides), were selected as acupoints protocol.BL30 is located on either side of the sacrococcygeal joint, approximately 1 cm from the joint. BL35 is in the buttock region, 0.5 cun lateral to the extremity of the coccyx.
  Interventions: Device: electroacupuncture
- conventional electroacupuncture (Active Comparator): The participants in the conventional electroacupuncture group will select RN3 (Zhongji), CV4 (Guanyuan), and ST28 (Shuidao, both sides), KL3 (Taixi).A needle measuring 0.25×40 mm will be inserted perpendicularly to a depth of 25- 40 mm to RN3, CV4 and ST28 and 0.5 cun to KL3 to induce a local sensation (distention or sourness).Subsequently, the electrodes from the SDZ-IIB electroacupuncture device will be connected to the needles at these points, with the anode connected to ST28 and RN3, the cathode connected to ST28 and CV4. The protocol includes the same duration, frequency of sessions and the parameter setting of electroacupuncture as for the'four sacral points'treatment.
  Interventions: Device: electroacupuncture

INTERVENTIONS:
Device: electroacupuncture — For'four sacral points'group, Hua Tuo brand disposable acupuncture needles (size 0.40 × 100mm) and electronic needle therapy instrument SDZ-IIB will be used.Bilateral BL30 and BL35, were selected as acupoints protocol.
  'Four sacral points'group consists of 8 sessions over an 4-week period after baseline(2 sessions in each week), each for 30minutes. The electroacupuncture will be set at a frequency of 2.0 Hz, continuous wave, a moderate intensity the patient can tolerate and 30 min during each treatment.
  Other Names: Acupuncture

SUMMARY:
Benign prostatic hyperplasia (BPH) is a common condition in aging men that is frequently associated with troublesome lower urinary tract symptoms (LUTS) which can be divided into storage phase symptoms (urinary frequency, urinary urgency, increased nocturia, urinary incontinence, etc.), voiding phase symptoms (interruption of urination, thinning of the urine line, straining to urinate, etc.), and post-void symptoms (incomplete sensation of urination, dribbling after urination, etc.).BPH is prevalent in as many as 40% of men in their fifties and 90% of men in their eighties.Yet, few effective therapiesare available for treating BPH/LUTS.

Acupuncture may be an effective treatment option for BPH/LUTS.However, effects of acupuncture on BPH/LUTS remain uncertain because of the small sample sizes or other methodological limitations.

The objective of this randomized,conventional electroacupuncture-controlled trial is to assess the effectiveness of electroacupuncture at'four sacral points'for relieving symptoms of BPH/LUTS. The results will provide a robust conclusion with a highlevel of evidence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPH in accordance with the criteria of the Chinese Urological Diagnosis and Treatment Guidelines 2014 edition.
* Male patients aged 40-80 years.
* Not on any 5a-reductase inhibitor, a1 receptor blocker or traditional Chinese medicine in the past two weeks.
* International Prostate Symptom Score (IPSS) scores range from 1 to 19.
* Family members or patients give informed consent and sign informed consent.

Exclusion Criteria:

* Patients with recurrent urinary tract infections.
* Patients with neurogenic bladder and urethral stricture, bladder tumor and prostate cancer.
* Patients with benign prostatic obstruction who have failed invasive treatment.
* Patients with serious cardiovascular and cerebrovascular diseases, hematopoietic system and other primary diseases and mental disorders.
* Patients who are participating in other clinical trials or who are participating in other clinical trials within one month.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
the Change From Baseline in the International Prostate Symptom Score (IPSS) | week4; week 8
  IPSS is a valid, reliable and sensitive measure for patients with lower urinary tract symptoms; it iswidely used in clinical practice and research to determine the severity of lower urinary tractsymptoms, including incomplete bladder emptying, frequency of urination, intermittency, urgency,weak urine stream, straining and nocturia. Each of the questions is rated from 0 (not at all) to 5(almost always). IPSS score ranges from 0 to 35, with higher score indicating more severe urinary symptoms.Significant effect was defined as most of the major symptoms and signs disappeared, and the score decreased between 60% and 89%.
  Effective is that the main symptoms and signs disappear partially, and the score decreases by 30%-59%.

SECONDARY OUTCOMES:
the Change From Baseline in the Overactive Bladder Symptom Score(OABSS) | week4; week 8
  OABSS is a valid self-assessment questionnaire, four questions were set according to OAB syndrome to determine the severity of OAB, which include daytime and nighttime urination frequency, urgency, urge incontinence. Score range is 0-15, with higher scores indicating increasing symptom severity.
the Change From Baseline in the Quality of Life Score(QOL) | week4; week 8
  The QOL score understands the subjective perception of BPH patients about the impact of their current symptoms on their quality of life and is divided into 7 levels, corresponding to a score of 0-6, with the higher the score the lower the patient's quality of life, mainly indicating the extent to which the patient suffers from LUTS.
the Change From Baseline in the Prostate Volume(PV) | week4; week 8
  Transabdominal urinary system B ultrasound examination, can understand whether the upper urinary tract water, expansion, prostate size, shape, whether hyperplastic glands burst into the bladder, the extent of burst, burst range, whether there is abnormal nodular echo, etc.. Then the anterior and posterior diameters, left and right diameters and upper and lower diameters of the prostate were measured respectively, and then the prostate volume was calculated according to the formula.
the Change From Baseline in the Post-Void Residual(PVR) | week4; week 8
  The measurement of PVR is basically the same as that of prostate volume. The three data of anterior and posterior diameters, upper and lower diameters and left and right diameters of residual urine were measured, and the residual urine volume was calculated according to the formula.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhou, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Result] Abrams P. Surgical Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: AUA Guideline Amendment 2020. Letter. J Urol. 2021 Mar;205(3):938. doi: 10.1097/JU.0000000000001558. Epub 2020 Dec 14. No abstract available. PMID 33315535